CLINICAL TRIAL: NCT04019535
Title: Diastolic Hyperemia Free Index for Assessment of Moderate Coronary Stenoses
Acronym: DFRiFR
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 201810120
Record Dates: First submitted 2019-03-29; First posted 2019-07-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: Physiologic assessment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: physiological assessment with Volcano Verrata pressure wire (iFR) — physiological assessment of the coronary lesion will be made with both iFR and dFR. all clinical decisions will be made based on the results of iFR
  Other Names: physiological assessment with Boston Scientific Comet pressure wire (dFR)

SUMMARY:
A total of 106 subjects will be enrolled at up to 3 sites. Initial enrollment will occur at Washington University only. After 15 subjects have been enrolled at the primary site and no serious adverse events or protocol events have occurred the additional sites will be trained and added to enrollment.

DETAILED DESCRIPTION:
With the release of DEFINE-FLAIR and iFR SWEDEHEART, coronary physiology and namely iFR, have robust clinical data supporting its routine use in the cardiac catheterization lab. Unfortunately, iFR is a proprietary algorithm owned by Phillips Volcano Corporation (San diego, California, USA) limiting the use of iFR to those centers with Volcano hardware. Whole cardiac cycle Pd/Pa has been another resting measure that has been evaluated and generally performs poorly compared to FFR. Although iFR is measured during the wave free period in diastole, to date there has been no assessment of diastolic Pd/Pa measurements and its potential correlation with the severity of coronary stenoses. Most importantly, evaluating the pressure differential across the entirety of diastole must by definition contain the "iFR value" and therefore should correlate very close with the iFR assessment. Preliminary unpublished data analyzing physiologic data in benchtop modeling from the VERIFY and CONTRAST studies suggest a very high correlation between iFR and diastolic Pd/Pa. This relationship strengthens when measurements are limited to 65% of diastole, hereby named the Diastolic hyperemia-Free Ratio (DFR). These data strongly suggest that DFR could be used as surrogate for iFR when iFR is not available and thus leverage the large clinical outcomes data for iFR in a new measure that is widely available to all standard coronary pressure wires.

Although this preliminary data is strong, none of these measures where made prospectively in actual patients and the iFR was measured off simulated benchtop pressure waveform modeling. This study aims to perform a real-time correlation and agreement between iFR and DFR in patients with moderate coronary stenoses and indications for physiologic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate Coronary lesion deemed to need iFR assessment - Angiographic severity of 40-70% that operator feels needs physiologic assessment
* Age 18-90 year old
* Single worst lesion per patient- Patients may have more than one lesion assessed but only 1 lesion will be evaluated per patient in this study

Exclusion Criteria:

* STEMI- Angiographic severity of 40-70% that operator feels needs physiologic assessment in setting of STEMI or 48hours within STEMI
* Atrial fibrillation
* Inability to provide informed consent- No surrogate or healthcare proxy will be allowed to consent for this study
* Severe tortuosity- Vessel tortuosity that the operator feels would be difficult to pass 2 pressure wires down or where pseudo lesions may be formed.
* Saphenous Vein Graft Lesion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate Coronary lesion deemed to need iFR assessment - Angiographic severity of 40-70% that operator feels needs physiologic assessment
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of iFR and DFR | The correlation between values will be the primary endpoint measured and occurs only during the index procedure.
  . DFR will be correlated, in VIVO, with the gold standard, diastolic coronary blood flow measurement, the instantaneous wave free ratio (iFR). Both DFR and iFR will be correlated simultaneously during the index procedure in patients with moderate coronary stenoses whom hemodynamic assessment was clinically indicated.
Agreement for treatment with iFR | after all subjects are enrolled the RedCap data will be evaluated
  . how many patients would be treated differently using iFR vs. DFR

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sintek, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided